CLINICAL TRIAL: NCT01207089
Title: A Phase I, Single Centre, Single-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD8329 After Administration of Multiple Ascending Doses in Abdominally Obese But Otherwise Healthy Male Subjects
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Administration of AZD8329
Acronym: AZ8329
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D2350C00010
Record Dates: First submitted 2010-09-14; First posted 2010-09-22 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Overweight; Healthy; Male
Keywords: Safety; tolerability; PK; healthy; overweight; obese
MeSH Terms: conditions — Overweight; Obesity | interventions — 4-(4-(2-adamantylcarbamoyl)-5-tert-butyl-pyrazol-1-yl)benzoic acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): AZD8329
  Interventions: Drug: AZD8329

INTERVENTIONS:
Drug: AZD8329 — AZD8329 Oral Solution 20mg/ml
  Arms: 2
Drug: Placebo — Placebo AZD8329 Oral Solution
  Arms: 1

SUMMARY:
The purpose of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD8329 following multiple ascending dose administrations in in overweight to obese but otherwise healthy male subjects.

DETAILED DESCRIPTION:
A Phase I, Single Centre, Single-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of oral AZD8329 after Administration of Multiple Ascending Doses in Abdominally Obese but otherwise Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 27 and 35 kg/m2 and a waist circumference greater than or equal to 102cm.
* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male subjects aged =20 to =50 years with suitable veins for cannulation or repeated venepuncture

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate.
* Fasting serum (S)-glucose =7.0 mmol/L or non-fasting S-glucose =11.1 mmol/L at screening.
* Any eating disorder or actively attempting to loose weight within 3 months prior to enrolment

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events). | Adverse events day -1
Safety variables (adverse events). | Adverse events will colletected entire study
Safety variables (clinical laboratory assessments). | Clinical labs day 1
Safety variables (clinical laboratory assessments). | Day 4
Safety variables (clinical laboratory assessments). | Day 8
Safety variables (clinical laboratory assessments). | Day 12
Safety variables (clinical laboratory assessments). | Clinical labs at follow up
Safety variables (adverse events) | Adverse events will colletected entire study
Safety variables (vital signs) | vital signs every hour during day 1
Safety variables (physical examination) | performed at screening
Safety variables (vital signs) | Vital Signs every hr during day 12
Safety variables (physical examination) | Performed at follow up
Safety variables (telemetry) | telemetry for 24hr. post dose day 1
Safety variables (telemetry) | telemetry for 24hr. post dose day 12
Safety variables (digital electrocardiograms (dECGs)) | dECG during 5min, 13 times 24 hr after dose day 1
Safety variables (digital electrocardiograms (dECGs)) | dECG during 5min, 13 times 24 hr after dose day 12
Safety variables (safety 12-lead paper electrocardiograms (pECG)) | pECG at screening
Safety variables (safety 12-lead paper electrocardiograms (pECG)) | pECG at follow up
Safety variables (clinical laboratory assessments). | clinical labs at screening
Safety variables (clinical laboratory assessments). | clinical labs day -3

SECONDARY OUTCOMES:
Pharmacokinetics Plasma and urine concentrations of AZD8329 and plasma and urine pharmacokinetics parameters | Information will be collected during day -1, day 1, 2, 3 and 12
Pharmacodynamic 11-βHSD1 enzyme activity in adipose tissue | Information will be collected from the time of day -1 throuout the study
Pharmacodynamic 11-βHSD1 enzyme activity in the liver by measuring prednisolone generation | Information will be collected from day -1 to follow up
To assess the effect on insulin after multiple doses of AZD8329 | Information will be collected from day -2 to follow up
To assess the effect on glucose after multiple doses of AZD8329 | Information will be collected from day -2 to follow up
To assess the effect on lipid variables after multiple doses of AZD8329 | Information will be collected from day -2 to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jan Eriksson, Study Chair — AstraZeneca; Dr. Mirjana Kujacic, Study Director — AstraZeneca; Dr. James Ritter, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Morentin Gutierrez P, Gyte A, deSchoolmeester J, Ceuppens P, Swales J, Stacey C, Eriksson JW, Sjostrand M, Nilsson C, Leighton B. Continuous inhibition of 11beta-hydroxysteroid dehydrogenase type I in adipose tissue leads to tachyphylaxis in humans and rats but not in mice. Br J Pharmacol. 2015 Oct;172(20):4806-16. doi: 10.1111/bph.13251. Epub 2015 Oct 8. PMID 26218540